CLINICAL TRIAL: NCT00341042
Title: Establishment of Normal Parameters for Blood and Sputum With Samples Obtained From Volunteers in Bamako
Brief Title: Collection of Tissue Specimens in Mali, West Africa, for HIV and Tuberculosis Research
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905028; 05-I-N028
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-05-01

CONDITIONS: Tuberculosis; HIV
Keywords: Normal Values; Complete Blood Count; HIV; Tuberculosis; Flow Cytometry
MeSH Terms: conditions — Tuberculosis

SUMMARY:
This study, conducted in Bamako, Mali (West Africa), will collect blood and sputum samples to establish normal values for laboratory test results among Malians. Researchers are starting a new initiative to study HIV and tuberculosis in Africa, using Mali as a model country. In order to perform these studies, the scientists need to know what constitutes normal laboratory values among the population. People in developing countries may have dramatically different laboratory values from those who live in developed countries, and there is currently little information available to distinguish normal from abnormal results in Malians. This study will establish normal ranges that will provide a basis for future HIV and tuberculosis research in Mali. Additionally it will provide blood and sputum samples to researchers to study different scientific questions related to HIV and Tuberculosis infection.

Healthy volunteers and people infected with HIV or tuberculosis, or both, who are 18 years of age or older and who live in Bamako, Mali, may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood test.

Participants provide a blood or sputum sample, or both, for laboratory analysis. Blood is collected through a needle inserted into an arm vein, and sputum is collected by having the participant cough deeply and spit in a cup. Participants may agree to provide samples one time only or on a returning visit basis. Returning visits may be scheduled daily or weekly. Subjects may continue to participate for the duration of the 4-year study, provided their medical history and physical examination are updated once a year.

DETAILED DESCRIPTION:
HIV and tuberculosis are major health issues in the developing world - HIV and tuberculosis affect several million people worldwide. Individually and together these two diseases kill more people than any other infections, with the worst suffering occurring on the African continent. Mali is a West African state awakening to the reality of these issues. While tuberculosis has always been a major problem in Mali, more recently HIV incidence has begun to increase.

We are commencing a new research initiative to study HIV and tuberculosis in Africa, using Mali as a model country. However, there is little baseline epidemiological, hematological, immunological or microbiological data to help distinguish normal from abnormal results; establishing normal population baseline values is necessary to facilitate future research. We will collect whole blood and sputum samples to establish baseline values, for the purpose of facilitating ongoing or future HIV and tuberculosis research. Specifically, samples will be used to determine normal hematological, immunological and other parameters for Malian people. In addition, we will use samples to optimize routine and specialized research assays. Sputum samples will be used in bacteriological and genetic studies intended to optimize studies relating to tuberculosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 yrs or older.

Adequate venous access.

Willingness to allow blood samples to be stored and used for future studies of HIV infection and pathogenesis.

Ability to sign informed consent and willingness to comply with study requirements and procedures.

EXCLUSION CRITERIA:

Anemia (Hg less than10 g/dl) (for patients donating blood only).

Underlying heart disease or bleeding disorder which in the judgment of the PI could increase the risk to the volunteer.

Fever of 101 degrees F or evidence of an acute infection. (for patients donating blood only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2005-01-04; Study Completion 2013-05-01

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Universite of Bamako, Bamako, Mali